CLINICAL TRIAL: NCT07009990
Title: The Greifswald Heart and Brain Project: Coronary and Cerebral Microvascular Dysfunction in Patients With Acute Neurological Diseases
Brief Title: Coronary and Cerebral Microvascular Dysfunction in Neurological Diseases
Acronym: G-HeBra
Status: Not yet recruiting | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: Department of Internal Medicine B, University Medicine Greifswald (Unknown); Institute for Diagnostic Radiology and Neuroradiology University Medicine Greifswald (Unknown); Department of Internal Medicine, First Clinic of Internal Medicine, University of Genoa, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: G-HeBra
Record Dates: First submitted 2025-05-19; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Epilepsy; Transient Global Amnesia (TGA)
Keywords: neurological diseases; cardiovascular health; perfusion; microvascular dysfunction; magnetic resonance imaging; transthoracic echocardiogram; cognitive function; stroke; transient global amnesia; epilepsy; brain health; microcirculation; Takotsubo syndrome
MeSH Terms: conditions — Stroke; Epilepsy; Amnesia, Transient Global; Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples (whole blood, serum, plasma)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Stroke patients: Patients who were referred to hospital due to an acute first-time stroke (ischemic or hemorrhage)
- Epilepsy patients: Patients who were referred to hospital due to an first-time generalized epileptic seizure (with focal or generalized onset)
- Transient global amnesia patients: Patients who were referred to hospital due to a transient global amnesia
- Control group for stroke patients: Participants who were recruited from data repositories of young and older participants without pre-existing neurological disease who had agreed to be re-contacted for future studies; will match the patient group with acute first-time stroke in terms of age, sex, hypertension, diabetes and smoking
- Control group for epilepsy and transient global amnesia patients: Participants who were recruited from data repositories of young and older participants without pre-existing neurological disease who had agreed to be re-contacted for future studies; will match the patient group with acute first-time generalized epileptic seizure and transient global amnesia in terms of age and sex

SUMMARY:
Neurological and cardiovascular diseases are increasing in relative and absolute terms globally, and pose a major burden in terms of morbidity, mortality, quality of life and healthcare costs. Increasing evidence has been found that disorders of blood circulation in the smallest vessels of the heart and the brain share similar risk factors as well as mechanisms but evidence about the potential link between both remains scarce.

Therefore, this study wants to investigate whether in patients with acute first-time stroke, first-time generalized epileptic seizure or first-time transient global amnesia, impairment in microcirculation is found in the brain and in the heart within 72 hours after the onset of first symptoms. We also intend to examine differences in structural brain as well as cardiac health parameters and in blood biomarkers between patients with acute neurological diseases and healthy controls matched for age, sex and major cardiovascular risk factors like diabetes, smoking and high blood pressure. In addition, we will characterize the cohorts in terms of cognitive function and questionnaires on lifestyle and self-reported emotional functioning. We expect lower circulation in the smallest blood vessels in the brain and in the heart in patients with acute neurological diseases compared to healthy controls.

This pilot project is intended to demonstrate feasibility and initial results and thus serve as the basis for a larger clinical trial to improve long-term cerebral and cardiac health in patients with acute neurological diseases

DETAILED DESCRIPTION:
Neurological and cardiovascular diseases are increasing in relative and absolute terms globally, and pose a major burden in terms of morbidity, mortality, quality of life and healthcare costs. Increasing evidence that microvascular dysfunction of the heart and the brain share similar disease risk factors as well as underlying pathophysiological mechanisms has been found but evidence about the potential link between both pathological processes is scarce.

This observational study will investigate whether in patients with acute neurological diseases (i.e., first-time acute stroke, first-time generalized epileptic seizure, or transient global amnesia [TGA]) without clinical evidence of acute coronary syndrome, microvascular dysfunction is found in the brain and in the heart within 72 hours (for TGA 24-72 hours) after onset of first symptoms.

A total of 60 in-patients who were referred to hospital due to an acute neurological disease including acute first-time stroke (ischemic or hemorrhage; N = 20), first-time generalized epileptic seizure (with focal or generalized onset; N = 20) and TGA (N = 20), will be included in the study. In parallel, two control groups of 20 individuals each will be recruited from data repositories of young and older participants without pre-existing neurological disease who had agreed to be re-contacted for future studies. One control group will match the patient group with acute first-time stroke in terms of age, sex, hypertension, diabetes and smoking. The other control group will match the patient groups with acute first-time generalized epileptic seizure and TGA in terms of age and sex.

Participants will be found in the University Medicine Greifswald, Department of Neurology, admitted to hospital due to an acute neurological event (i.e., first-time acute stroke, first-time generalized epileptic seizure, or TGA). The G-HeBra study team from Neurology will check daily with the Neurologist on call for new hospitalizations due to the aforementioned acute neurological events and those patients will be visited as soon as possible by the G-HeBra study team; to be informed about the study. The G-HeBra study team will ascertain inclusion and exclusion criteria with the patient. If the patient is suitable and willing to participate in the study after receiving both oral and written information, the patient will sign the informed consent. After giving written informed consent, an identification number will be assigned for pseudonymization. Informed consent may be revoked at any time without any reason.

Appointments for the different study assessments will be made within 72 hours (for TGA after 24 hours up to 72 hours) after onset of first symptoms. The collection of demographic data, neuropsychological tests, questionnaires and a standardized medical examination including blood sampling will be conducted during the same visit, if possible. Further visits will be scheduled for cerebral and cardiac magnetic resonance imaging (MRI), transthoracic echocardiography (TTE) with strain, measurement of microvascular endothelial function, and angiography-derived assessment of coronary microvascular function. All assessments will be conducted as early as possible after the acute neurological event.

In parallel, the G-HeBra study team will contact individuals for the control group from data repositories by telephone and interview them to decide whether or not they may be included in the study. If a person fulfills the in- and exclusion criteria, the G-HeBra-study team will collect biographical and general information about the participant and will provide first information about the study procedure. Participants of the control group will also have all assessments at the University Medicine Greifswald, starting with oral and written informed consent. After giving written informed consent, an identification number will be assigned for pseudonymization and informed content may be also revoked at any time without any reason.

On-site, for all participants, the examiner will first collect biographical and general information about the participant and will give detailed information about the study procedure. A medical assessment including an interview on own's medical history as well as on family history, standardized medical examination and collection of anthropometric data will be conducted. For comparability, blood collection will take place in the morning (between 6am and 11am) for all participants and within 24 hours after study enrollment for hospitalized patients. Pre-analytics for the basic laboratory and the differential blood analysis are carried out according to established standard instructions. The total blood volume in this study is 35.7 ml and will be collected during one blood draw.

Cognitive and neuropsychological assessment will include the Mini Mental State Examination and further tests for assessing verbal memory, object recognition memory, working memory, executive functions, and attention. Premorbid intelligence quotient is tested as well as questionnaires on depressive symptoms, stress coping, lifestyle and cardiac health will be completed.

Cerebral and cardiac MRI will take place in one session at the University Medicine Greifswald and will not exceed 60 minutes. Scanning will be conducted on a 3-Tesla Siemens MR-systems at the Department of Radiology, University Medicine Greifswald. Participants will be interviewed for MRI contraindications prior to study enrollment and will be excluded from study participation if one of the exclusion criteria applies.

The cerebral MRI will include structural and functional/perfusion sequences using a 64-channel head coil. Perfusion brain images will be acquired using a pseudo-continuous-arterial spin labeling sequence for cerebral blood flow quantification during rest. T1-weighted three-dimensional magnetization-prepared rapid acquisition gradient echo images will be acquired to evaluate structural brain features, such as cortical thickness, cortical surface area and cortical/subcortical volume of brain regions of interest. Fluid attenuated inversion recovery T2-weighted images will be acquired to detect white matter hyperintensities and microbleeds.The MRI images will be analyzed using standard procedures and software packages, for example SPM (Welcome Department of Imaging Neuroscience, University College London, UK) and Matlab (Mathworks, Sherborn, Massachusetts, USA), VBM toolbox (Structural Brain Mapping Group, University of Jena, Germany), SPSS (SPSS Inc., Chicago, Illinois, USA), FMRIB Software Library (FSL; http://www.fmrib.ox.ac.uk/fsl), and FreeSurfer. Cardiac MRI will incorporate both standard and advanced imaging sequences. Cine sequences will assess cardiac contractile function. Advanced techniques including myocardial perfusion reserve, myocardial blood flow, native T2, native and post-contrast T1 mapping, intravoxel incoherent motion, perfusion MRI, and including index of microcirculatory resistance will enable a comprehensive evaluation of myocardial function, tissue characteristics, and coronary microvascular function. Gadolinium-based contrast agents will be used for late gadolinium enhancement, which is essential to detect myocardial scarring, fibrosis, and previous infarctions.

TTE with strain, measurement of microvascular endothelial function, and angiography-derived assessment of coronary microvascular function will take place at the Department of Internal Medicine B, University Medicine Greifswald, Germany, and takes about 60 minutes. Echocardiography as a non-invasive gold standard for determining left and right ventricular function and morphology as well as assessing valve function (Vingmed Vivid 9, 5S transducer 2.0 - 5.0 megahertz, GE Medical Systems GmbH, Hamburg, Germany) will be performed and assessed by two expert operators. Measurements will include left ventricular ejection fraction for systolic function, global longitudinal strain for myocardial deformation, and left atrial strain for atrial function. For diastolic function, parameters will include the E/A ratio, E/e' ratio, left atrial volume index, deceleration time of the mitral inflow, and isovolumetric relaxation time. Additionally, right ventricular systolic function and pulmonary pressures will be assessed using tricuspid annular plane systolic excursion, fractional area change, and systolic pulmonary arterial pressure, estimated from tricuspid regurgitation velocity and right atrial pressure.

Endothelial function will be assessed using the EndoPAT device (Itamar Medical Ltd., Israel), a plethysmographic method that employs pneumatic finger sensors. The procedure begins after a resting phase of at least 5 minutes in a lying position to ensure stable baseline conditions. The blood flow in the right index finger is continuously monitored. Following the baseline measurement, a blood pressure cuff is inflated to 220 mmHg on the upper arm for 5 minutes to induce temporary occlusion of blood flow. After deflating the cuff, blood flow is measured again for one minute to evaluate the post-occlusive reactive hyperemia response, which reflects endothelial function. The EndoPAT device calculates the Reactive Hyperemia Index, which is a measure of endothelial function.

The angiography-derived assessment of coronary microvascular function provides a non-invasive method for evaluating coronary resistance and microvascular health without the need for a coronary wire. Parameters such as μFR (microvascular Fractional Reserve) and AMR (Angio-based Microvascular Resistance) are derived from 2D or 3D reconstruction and fluid dynamic analysis of standard angiographic images. μFR offers physiological assessment of both main vessels and side branches, while AMR allows for the efficient identification of microvascular dysfunction without additional procedural risks. This assessment will be calculated in the subgroup of patients undergoing coronary angiography for clinical indications.

Regarding statistical analyses, we will first descriptively evaluate the prevalence of acute neurological patients (stroke, epileptic seizure, TGA) with microvascular dysfunction in the brain and heart in our study sample. The primary outcome will be statistically analyzed for each patient group (stroke, epileptic seizure, TGA) and the corresponding control group separately using linear mixed models with microvascular function in the brain/heart as dependent variable and group (patient or control) as independent variable adjusted for age and sex including random intercept for the matching identification number. In terms of secondary outcomes, we will evaluate differences in blood biomarkers, cerebral structural measures, additional cardiac parameters from MRI and TTE, and microvascular endothelial function parameters between the patient groups and the corresponding control groups using linear mixed models adjusted for age and sex including random intercept for the matching identification number. Moreover, multiple linear regression models will be conducted to analyze the association between cerebral (as well as coronary) microvascular dysfunction (dependent variable) and our secondary outcome measures (e.g., blood biomarkers, cerebral structural measures, additional cardiac parameters from MRI and TTE, and parameters of microvascular endothelial function; independent variable) in each patient group with acute neurological event separately. In addition, all participants will be characterized descriptively and by using linear mixed models in terms of cognitive performance and by evaluating questionnaires on lifestyle and emotional functioning. As these are all exploratory analyses (non confirmatory) in this study, we will rather focus on estimating effect sizes (e.g., Cohen's d or Cohen's f) than on statistical significance in our models.

This pilot project is intended to demonstrate feasibility and initial results and thus serve as the basis for a possible larger clinical trial to improve long-term cerebral and cardiac health in patients with acute neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, minimum age: 45 years
* Gave informed consent
* Specifically for patient group: Admission to hospital due to an acute neurological event due to acute first-time stroke (ischemic or hemorrhage; mild to moderate in severity based on The National Institutes of Health Stroke Scale [NIHSS], score <15) and able to provide informed consent (e.g., no or only mild aphasia; no impairment of consciousness), first-time generalized epileptic seizure (with focal or generalized onset), or transient global amnesia

Exclusion Criteria:

* History of stroke or any type of seizure
* Neurodegenerative neurological disorders including dementia, Parkinson's disease, Huntington's disease, and Amyotrophic lateral sclerosis
* Acute myocardial infarction requiring revascularization
* Severe and untreated medical conditions, including advanced-stage malignant tumors and cardiac diseases resulting in cardiogenic shock or acute heart failure
* Severe infections (C-Reactive Protein [CRP] > 50 mg/dL)
* History of severe alcoholism or use of drugs
* Severe psychiatric disorders such as moderate to severe depression (if not in remission) or psychosis
* Contraindication to magnetic resonance imaging or renal dysfunction with eGFR (estimated glomerular filtration rate) < 30 ml/min/1.73 m2, which would not allow the administration of the contrast agent gadolinium

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted with acute neurological event to the University Medicine Greifswald and healthy controls from the general population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Microvascular function in the brain and heart | at Baseline
  For the brain, this will involve quantification of cerebral blood flow in the whole brain using arterial spin labeling magnetic resonance imaging technique.
  The cardiac microvascular function will be evaluated primarily through the measurement of coronary flow reserve with cardiac magnetic resonance imaging.

SECONDARY OUTCOMES:
Cerebral MRI | at Baseline
  Cerebral structural measures (e.g. grey matter atrophy, white matter lesions), operationalized by different magnetic resonance imaging techniques including T1-weighted magnetization-prepared rapid acquisition gradient echo and fluid attenuated inversion recovery
Cardiac MRI | at Baseline
  Analysis of myocardial perfusion reserve, myocardial blood flow, cine sequences, intravoxel incoherent motion, extracellular volume fraction and gadolinium enhancement to assess both functional and structural aspects of cardiac microvascular health and tissue characteristics
Cardiac function and myocardial deformation | at Baseline
  Transthoracic echocardiography parameters, including left ventricular systolic and diastolic function, global longitudinal strain, left atrial strain and right ventricular systolic function
Microvascular endothelial function and coronary microvascular dysfunction | at Baseline
  Microvascular endothelial function: non-invasively assessed by EndoPAT, a device that measures endothelial health through peripheral arterial tonometry.
  Coronary microvascular dysfunction: assessed with angiography-derived methods in form of index of microcirculatory resistance and coronary flow reserve. Only in patients undergoing coronary angiography due to a clinical indication.
Blood Biomarkers related to heart function | at Baseline
  Measuring of blood biomarkers related to heart function
Blood Biomarkers related to endothelial dysfunction | at Baseline
  Measuring of blood biomarkers related to endothelial dysfunction
Blood Biomarkers related to brain injury | at baseline
  Measuring of blood biomarkers related to brain injury
Blood Biomarkers related to stress | at Baseline
  Measuring of blood biomarkers related to stress
Blood Biomarkers related to general health | at Baseline
  Measuring of blood biomarkers related to general health

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof. Dr., Principal Investigator — University Medicine Greifswald; Christian Templin, Prof. Dr. Dr., Principal Investigator — University Medicine Greifswald; Claudia Schwarz, Dr., Principal Investigator — University Medicine Greifswald; Davide Di Vece, Dr., Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No